CLINICAL TRIAL: NCT00107887
Title: Impact of TB Preventive Therapy for HIV/TB Co-infected Patients With Access to Highly Active Antiretroviral Therapy in Rio de Janeiro, Brazil: A Phased Implementation Trial
Brief Title: TB (Tuberculosis) Preventive Therapy for HIV Patients With Access to HAART (Highly Active Antiretroviral Therapy)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Consortium to Respond Effectively to the AIDS/Tuberculosis Epidemic (Other); Communicable Disease Program, Brazil (Other Government); Bill and Melinda Gates Foundation (Other)
Responsible Party: Dr. Richard Chaisson, Center for Tuberculosis Research, Johns Hopkins University
Organization: Communicable Disease Program, Brazil (Other Government)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 19790.01
Record Dates: First submitted 2005-04-11; First posted 2005-04-12 (Estimated); Last update posted 2011-06-15 (Estimated); Status verified 2011-06

CONDITIONS: Tuberculosis; HIV Infections
Keywords: TST; isoniazid; HAART; Brazil; HIV
MeSH Terms: conditions — Tuberculosis; HIV Infections | interventions — Tuberculin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (No Intervention): Subjects in clinics that have not received the intervention
- 2 (Experimental): Subjects at clinics that have received the intervention
  Interventions: Drug: INH preventive therapy; Drug: TST (tuberculin skin test)

INTERVENTIONS:
Drug: INH preventive therapy — Clinics will receive training regarding the use of IPT for prevention of Tuberculosis
  Arms: 2
Drug: TST (tuberculin skin test) — Clinics will be trained in the use of TST for assessing exposure to TB
  Arms: 2

SUMMARY:
The purpose of this study is to determine if implementing a policy of widespread INH (Isoniazid) prophylaxis therapy in HIV-infected patients with access to antiretroviral therapy reduces the incidence of active TB disease in the HIV clinic population.

DETAILED DESCRIPTION:
Tuberculosis remains a major public health problem in Brazil. Approximately 35% of HIV-infected adults in Rio de Janeiro are co-infected with latent TB. The Brazilian policies for the provision of treatment to HIV-infected people are among the most progressive in the world. Brazil provides combination antiretroviral therapy free of charge to all patients who meet clinical criteria and maintains an extensive clinic and laboratory system for the appropriate prescription and monitoring of therapy. The use of IPT, however, has been very limited in Brazil and TB remains a prominent disease in AIDS patients.

A clustered randomized trial (CRT) will determine if the routine detection of latent TB in HIV-infected patients identified at HIV clinics in Rio de Janeiro, followed by treatment with isoniazid, will reduce TB incidence in this population. The CRT will take a phased-implementation approach to ensure that all clinics will eventually have full coverage.

This study will determine if implementing a policy of widespread IPT use in HIV-infected patients with access to ARV therapy reduces the incidence of active TB disease in the HIV clinic population. The study population will be comprised of HIV-infected individuals who attend any of the 29 government HIV clinics in Rio de Janeiro, Brazil. We expect that IPT use in addition to ARVs will result in a 40-60% reduction in TB incidence, and that approximately 50% of the prevented TB cases will be in patients not yet eligible for HAART.

ELIGIBILITY:
Inclusion Criteria:

* Attending 1 of 29 participating HIV clinics
* Confirmed HIV infection
* Age > 15 years

Exclusion Criteria:

* Current active TB disease
* TB infection within 2 years
* Hepatitis

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17415 (Actual)
Dates: Start 2005-06; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Measured incidence of active TB in HIV clinic population before and following implementation of IPT policy | 6 Years
Comparative impact of IPT (Isoniazid Preventive Therapy) and ARVs (antiretrovirals) on TB incidence in the HIV clinic population | 6 Years

SECONDARY OUTCOMES:
Characteristics of TST+ vs. TST+ HIV-infected patients | 6 Years
Clinical, demographic and laboratory predictors of developing active TB | 6 Years
Lessons learned related to training and implementation | 6 Years

CONTACTS AND LOCATIONS:
Overall Officials: Valeria Saraceni, MD, Study Director — City of Rio De Janeiro Municipal Health Secretariat; Richard E Chaisson, M.D., Principal Investigator — Johns Hopkins University; Betina Durovni, M.D., Study Chair — City of Rio de Janeiro Municipal Health Secretariat
Locations (1):
- City of Rio De Janeiro Health Department Clinics, Rio de Janeiro, Rio de Janeiro, Brazil

REFERENCES:
- [Background] Golub JE, Durovni B, King BS, Cavalacante SC, Pacheco AG, Moulton LH, Moore RD, Chaisson RE, Saraceni V. Recurrent tuberculosis in HIV-infected patients in Rio de Janeiro, Brazil. AIDS. 2008 Nov 30;22(18):2527-33. doi: 10.1097/QAD.0b013e328311ac4e. PMID 19005276
- [Background] Golub JE, Saraceni V, Cavalcante SC, Pacheco AG, Moulton LH, King BS, Efron A, Moore RD, Chaisson RE, Durovni B. The impact of antiretroviral therapy and isoniazid preventive therapy on tuberculosis incidence in HIV-infected patients in Rio de Janeiro, Brazil. AIDS. 2007 Jul 11;21(11):1441-8. doi: 10.1097/QAD.0b013e328216f441. PMID 17589190
- [Derived] Durovni B, Saraceni V, Moulton LH, Pacheco AG, Cavalcante SC, King BS, Cohn S, Efron A, Chaisson RE, Golub JE. Effect of improved tuberculosis screening and isoniazid preventive therapy on incidence of tuberculosis and death in patients with HIV in clinics in Rio de Janeiro, Brazil: a stepped wedge, cluster-randomised trial. Lancet Infect Dis. 2013 Oct;13(10):852-8. doi: 10.1016/S1473-3099(13)70187-7. Epub 2013 Aug 16. PMID 23954450
- See also: Related Info — http://www.tbhiv-create.org